CLINICAL TRIAL: NCT04940468
Title: Do Decreased Dietary Fat and Increased Fiber Reduce Recurrence of Clostridioides Difficile Infection in Oncology Patients?
Brief Title: High- Fiber/ Low-fat Diet for Prevention of Recurrent Clostridioides Difficile Infection in Oncology
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed by PI due to low accrual
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-2851.cc; P30CA046934 (NIH); U01AI150589-01A1 (NIH)
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Leukemia, Lymphocytic, Acute; Leukemia, Myeloid, Acute; Lymphoma; Clostridium Difficile Infection
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma; Clostridium Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Diet Intervention (Active Comparator): Based on participant food preferences, diet higher in fiber and lower in fat than the participant's typical diet will be provided.
  Interventions: Other: Diet Intervention
- Arm 2: No Diet Intervention (No Intervention): No diet changes will be made for participants

INTERVENTIONS:
Other: Diet Intervention — The dietary fiber intake target will be 19 g/d for ages 9-18 and females age 19 and older and 23g/d for males age 19 and older.
  Arms: Arm 1: Diet Intervention

SUMMARY:
The primary objective of the study is to determine whether dietary intervention to increase fiber and decrease fat reduces C. difficile infection recurrence in a cohort of oncology patients.

DETAILED DESCRIPTION:
This is a randomized study. A total of 124 individuals with either acute leukemia or lymphoma and a first or second occurrence of C. difficile infection will be enrolled. Participants will be randomized to Arm 1 (Diet intervention) or Arm 2 (No diet intervention). Participants in Arm 1 will be assessed for food preferences and will be provided lists of high fiber and high saturated fats. Participants will be able to choose foods from the high fiber food lists and groceries will be provided once per week to support each participant's meal plan. Participants will be asked to limit foods on the high saturated fats list. Food consumption with a 24 hour recall and weight will be monitored and stool samples will be collected one time per week for 6 weeks. In Arm 2, participants will be asked to provide 24 hour food recall and stool samples. Individuals in both arms will be monitored for stool consistency and any antibiotics or chemotherapy drugs taken. Participation will last 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a malignant neoplasm at the at Children's Hospital Colorado or the University of Colorado Hospital
* Diagnosis of first time or first recurrent CDI as defined by clinical criteria within the past 21 days
* Informed consent obtained and signed. For minors, the consent will be completed by a guardian and the study participant will sign the assent form. Only the consent form is required of adults.
* 9 years old or older
* 40th to 100th percentiles of saturated fat intake and below the 50th percentile for fiber intake based on a food frequency questionnaire.
* Ability to comply with study procedures for the entire length of the study.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2026-01-12 (Actual)

PRIMARY OUTCOMES:
C. difficile infection recurrence (yes/no) | 6 months
  Signs of active diarrhea using Bristol stool scale. The Bristol stool form scale includes seven types of stool which ranging from constipation (type 1) to diarrhea (type 7).

SECONDARY OUTCOMES:
C. difficile toxins A and B | 6 weeks
  Quantify toxins in stool using "Separate detection of C. difficile toxins A and B" kit (tgc Biomics)
Fecal microbiome | 6 weeks
  Characterize the microbiome in fecal samples as using 16S rRNA targeted and shotgun metagenomic sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lozupone, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Childrens Hospital Colorado, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No